CLINICAL TRIAL: NCT00614588
Title: Accuracy of Temperature Measurement in Post-Anesthesia Care Units
Brief Title: Temperature Measurement in Post-Anesthesia Care Units
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 07-986
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Surgery; Postoperative; Laparoscopic Surgery; General Anesthesia
Keywords: temperature; monitor; surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- observation group: Patients undergoing laparoscopic surgery requiring general anesthesia and a bladder catheter.
  Interventions: Device: Body temperature thermometers

INTERVENTIONS:
Device: Body temperature thermometers — Temperature readings every 30 minutes during and post surgery using internal stethoscope, catheter and adhesive patches/electronic thermometer.
  Other Names: 1. Distal esophagus (Mon-a-therm, Tyco-Mallinckrodt Anesthesia Products,; 2. Bladder (Mon-a-therm, Tyco-Mallinckrodt Anesthesia Products,; 3. Infrared-aural canal bilaterally (GENIUS Model 3000A, Kendall Healthcare); 4. Temporal artery with an electronic scanning thermometer (Model TAT-5000, Exergen); 5. Posterior sublingual pocket with electronic thermometer (Turbo Temperature Model 2180CX01EE); 6. Forehead skin thermocouple (Mon-a-therm, Tyco-Mallinckrodt Anesthesia Products); 7. Axilla with an electronic probe (Mon-a-therm, Tyco-Mallinckrodt Anesthesia Products); 8. Forehead liquid-crystal (Crystaline II); 9. Intermittent axillary temperature (Turbo Temperature Model 2180CX01EE); 10. "Deep" temperature with a 4-cm probe on the forehead; 11. "Deep" temperature with a 7-cm probe over the subclavicular region of the upper chest

SUMMARY:
This study will evaluate the accuracy of several thermometers and temperature changes during surgery and immediately after surgery.

DETAILED DESCRIPTION:
Several measurements of temperature will be taken at 30 minute intervals during surgery under general anesthesia and in the post operative care unit. Measurements will be taken as follows:

* esophagus using an internal stethoscope
* urinary bladder using a catheter
* ear canal
* skin of the forehead using adhesive devices(4 thermometers)
* axilla ("armpit") using adhesive devices(2 thermometers)
* mouth
* skin of the upper chest

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years of age
* American Society of Anesthesiologists (ASA) physical status of 1-3
* laparoscopic surgery of the abdomen or pelvis that is expected to require general endotracheal anesthesia and insertion of a Foley catheter expected to be in place for at least one hour after surgery

Exclusion Criteria:

* under 18 or over 80 years of age
* pre-existing nasogastric tube
* require bispectral index monitoring
* upper esophageal disease
* forehead rash or infection, oral infection or trauma, or ear infection or drainage

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing laparoscopic surgery requiring general anesthesia and a bladder catheter.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2008-01; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
To determine the accuracy of various temperature-monitoring methods and sites suitable for Post Anesthesia Care Unit use. | Discharge from Post Anesthesia Care Unit

SECONDARY OUTCOMES:
To quantify the core temperature changes that occur during transport from the Operating Room to the PostAnesthesia Care Unit. | PostAnesthesia Care Unit

CONTACTS AND LOCATIONS:
Overall Officials: Daniel I Sessler, MD, Study Chair — The Cleveland Clinic; Daniel I Sessler, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States